CLINICAL TRIAL: NCT05822674
Title: A Preliminary Clinical Study on the Effects of Oral Hypoglycemic Agents on the Stress Hyperglycemic Ratio in Type 2 Diabetes Patients in the Absence of Serious Illness
Brief Title: Variable Effects of Anti-diabetics on Stress Hyperglycemia Ratio
Status: Completed | Type: Observational
Sponsor: University of Diyala (Other)
Responsible Party: Principal Investigator, Marwan Salih Mohamad Al-Nimer, Emeritus Professor, University of Diyala
Other Study IDs: University of Diyala
Record Dates: First submitted 2023-03-08; First posted 2023-04-21 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Type 2 Diabetes
Keywords: Stress hyperglycemia ratio; Sitagliptin; Empagliflozin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate; Metformin; Tablets; empagliflozin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sitagliptin/metformin: Patients with T2D treated with sitagliptin/metformin (50/500mg) once daily for 10 weeks
  Interventions: Drug: Sitagliptin/metformin ( 50/500mg) Oral Tablet
- Empagliflozin/metformin: Patients with T2D treated with empagliflozin/metformin (10/500mg) once daily for 10 weeks
  Interventions: Drug: Empagliflozin/metformin(10/500mg) Oral Tablet

INTERVENTIONS:
Drug: Sitagliptin/metformin ( 50/500mg) Oral Tablet — The drug was prescribed once daily per oral for 10 weeks
  Other Names: Group I
  Groups: Sitagliptin/metformin
Drug: Empagliflozin/metformin(10/500mg) Oral Tablet — The drug was prescribed once daily per oral for 10 weeks
  Other Names: Group II
  Groups: Empagliflozin/metformin

SUMMARY:
A blood glucose level of equal to or greater than 180 mg/dL that occurred during stress in a patient without diabetes mellitus (DM) is termed stress hyperglycemia (SH). The stress hyperglycemia ratio (SHR) is defined as the fasting blood glucose divided by the blood glucose level that is calculated from the glycosylated hemoglobin (HBA1c) value on admission. A significantly higher SHR is associated with worse prognostic biomarkers in diabetic patients with complications

DETAILED DESCRIPTION:
Stress hyperglycemia (SH) is an increase in circulating glucose levels in biological fluids as a physiological response to stress in diabetic patients who are known or newly diagnosed, or a pathological condition associated with in-hospital-related hyperglycemia.

Interventions. Through their pleiotropic effects, some oral hypoglycemic agents improved stress hyperglycemia. When compared to non-SGLT-I (sodium glucose transporter-inhibitor) users, diabetic patients who used (SGLT-I) and had an acute myocardial infarction had less prevalent stress hyperglycemia, a smaller infarct size, and evidence of a low inflammatory response. The rationale this study is to evaluate the SHR in T2D patients who do not have serious illnesses and are managed with oral hypoglycemic agents

ELIGIBILITY:
Inclusion Criteria:

* Age ≥35 years
* Diagnosis of Type 2 diabetes
* Absence of serious illnesses
* No evidence of trauma

Exclusion Criteria:

* Overt complications of diabetes
* Any participant used antibiotics for infectious diseases
* Any participant used non-steroidal antiinflammatory drugs
* Current or past history of mental diseases
* Current hematological diseases
* Pregnancy
* Nursing mothers

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Known cases of type 2 diabetes who were attending the diabetes centers and private clinics seeking for diabetes control and follow-up.
  The authors discussed with the participants about the study design and outcomes
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Stress hyperglycemia Ratio | 10 week
  The ratio of stress-to-on admission blood glucose was calculated

SECONDARY OUTCOMES:
Hematological indices | 10 week
  Concentration of hemoglobin (g/dL) and the value of mean corpuscular volume (fL)
Inflammatory markers | 10 week
  Concentration of c-reactive protein (mg/L)

CONTACTS AND LOCATIONS:
Overall Officials: Ismail Latif, Study Director — The Dean College of Medicine, University of Diyal
Locations (1):
- College of Medicine, University of Diyala, Baqubah, Diyala Governorate, Iraq

IPD SHARING:
Plan to Share IPD: Undecided
The data of this study can be shared on request